CLINICAL TRIAL: NCT01264874
Title: Phase III, Randomized, Double Blind Trial on Vitamin D Supplementation for Resected Stage II Melanoma Patients
Brief Title: MelaViD: A Trial on Vitamin D Supplementation for Resected Stage II Melanoma Patients
Acronym: MelaViD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor accrual rate
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S480/209; 2009-012049-46 (EudraCT Number)
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2017-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (Experimental): Vitamin D3 administration
  Interventions: Drug: Vitamin D3 ( Colecalciferol)
- placebo (Placebo Comparator): matched placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Vitamin D3 ( Colecalciferol) — 100000 IU every 50 days for 3 years
  Other Names: dibase
  Arms: Vitamin D3
Other: placebo — For 3 years IU every 50 days
  Arms: placebo

SUMMARY:
The purpose of this trial is to assess the effect of vitamin D supplementation on recurrence in resected stage II melanoma patients.

DETAILED DESCRIPTION:
Cancer chemoprevention uses natural, synthetic, or biologic chemical agents to reverse, suppress, or prevent carcinogenic progression (Sporn MB Cancer Res 1976). Genetic changes exist throughout the field and increase the likelihood that one or more premalignant and malignant lesions may develop within that field. Multistep carcinogenesis describes a stepwise accumulation of alterations, both genotypic and phenotypic. Arresting one or several of the steps may impede or delay the development of cancer. Several epidemiological, pre-clinical and clinical studies support Vitamin D as preventive and therapeutic cancer agent, for a wide spectrum of cancer. Calcitriol (1,25-dihydroxyvitamin D [1,25(OH) D]), the hormonal derivative of vitamin D, has been established since the 1980s as an antiproliferative and prodifferentiation agent, and as a proapoptotic agent and an inhibitor of cell migration, which may imply an inhibitory effect in cancer. Vitamin D is more like a hormone and not strictly a vitamin according to the classical criteria that an essential nutrient is a substance the body cannot synthesise in sufficient quantities itself. Also, vitamins are usually involved in biochemical reactions, while 1_,25-dihydroxyvitamin D exerts its action via VDR. Vitamin D is a group of fat-soluble prohormones, the two major forms of which are vitamin D2 (or ergocalciferol) and vitamin D3 (or cholecalciferol). Endogenous synthesis of vitamin D3 takes place in the skin under the influence of ultra violet B (UVB) radiation. Exogenous vitamin D2 or D3 comes from dietary intake. The overall vitamin D intake is the sum of cutaneous vitamin D and nutritional vitamin D and D. Vitamin D on its own has no physiological action. To be physiologically active, vitamin D must first be hydroxylated in the liver by the enzyme 25-hydroxylase, encoded by CYP27A1 (also called the 25-hydroxylase) in 25-hydroxyvitamin D or 1,25-hydroxyvitamin D (1,25-hydroxyvitamin D). The 25-hydroxyvitamin D is inactive, and an additional hydroxylation in the kidney by the enzyme 1_-hydroxylase, encoded by CYP27B1, (also called 1_-hydroxylase) is necessary for production of the physiologically active vitamin D metabolite, the 1_,25-dihydroxyvitamin D (calcitriol). When 1,25(OH) D is sufficiently available, the enzyme mitochondrial protein encoded by CYP24A1 metabolises the 1_,25-dihydroxyvitamin D in 1_,24,25-dihydroxyvitamin D, which is further catabolised to calcitroic acid. 25(OH)D and 1,25(OH)2D are transported in serum by the vitamin D-binding protein (gene name: GC, group-specific component). Ahn systematically investigated the association of 48 SNPS in four vitamin D metabolizing genes (CYP27A1, GC, CYP27B1, and CYP24A1) with serum 25(OH)D levels. Four tagSNPS in GC, the major serum 25(OH)D carrier, were associated with 25(OH)D levels (Ahn et al.Carcinogenesis 2009). CYP24A1 encodes a member of the cytochrome P450 superfamily of enzymes. The cytochrome P450 proteins are monooxygenases which catalyze many reactions involved in drug metabolism and synthesis of cholesterol, steroids and other lipids. This mitochondrial protein initiates the degradation of 1,25-dihydroxyvitamin D by hydroxylation of the side chain. In regulating the level of vitamin D, this enzyme plays a role in calcium homeostasis and the vitamin D endocrine system. Of interest, epigenetic silencing of CYP24A1, which is overexpressed in many cancers, in tumour-derived endothelial cells renders the tumour sensitive to the anti-angiogenic effects of 1,25(OH) D. Various molecules can inhibit 24-Ohase. These merit exploration and further development as specific small molecule 24-OHase inhibitors, especially in combination with 1,25(OH)D or other vitamin D analogues. These may maximize intracellular 1,25(OH)D content and exert optimal antiproliferative effects (Deeb 2007; Mantell 2000; Nishimura 1994). Binding of 1,25(OH)D to the vitamin D receptor (VDR) suppresses proliferation and induces differentiation of cancer cells in tumour tissue, suggesting that high levels of vitamin D metabolites may be protective against cancer (Deeb 2007; Reichel 1989).

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old with newly diagnosed histologically proven resected melanoma
2. Stage: IIa (T2b, T3a), IIb (T3b T4a) and IIc (T4b), N0, M0
3. Signed informed Consent
4. Willingness to provide blood samples
5. Performance Status of 0-1
6. Hematopoietic functionality at the entry of the study: leukocytes, platelets, haemoglobin and neutrophiles within the normal limits of laboratory references
7. Hepatic and renal functionality at the entry of the study within the normal range of each laboratory
8. Serum and urinary calcium within the upper limit of laboratory references.

Exclusion Criteria:

1. Primary not cutaneous melanoma
2. Clinical/radiological evidence or laboratory/pathology report of not completely resected melanoma
3. History of cancer (other than Carcinoma in situ (CIN) and non melanoma skin cancere (NMSC)
4. Current daily use of at least 600 IU/day of supplemental vitamin D or calcitriol or high dose of calcium therapy (e.g. calcium citrate with vitamin D) within the prior 6 months greater than 600 mg calcium per day during study
5. History of recurrent renal calculi or hypercalcemia (>10mg/dl), current and chronic use of oral corticosteroids
6. History of malabsorption syndrome (e.g., pancreatic insufficiency, celiac disease, Crohn disease or tropical sprue)
7. History of small intestinal resection (e.g., ileal bypass surgery for treatment of morbid obesity resection > 50 % of slim bowel)
8. Hypersensitivity to cholecalciferol or one of its components
9. Chronic liver disease, chronic renal disease, or renal dialysis
10. History of parathyroid disease and sarcoidosis
11. Pregnancy or breast feeding or planning on becoming pregnant during the 3 years of treatment
12. Chronic alcoholism
13. Any medical condition that in the physician's opinion would potentially interfere with vitamin D absorption, such as celiac sprue, ulcerative colitis, patients treated pharmacologically for obesity
14. Any logistic condition that do not allow follow-up of the disease of the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Disease free survival and Overall Survival | 3 years of treatment and 2 of follow up
  Disease free survival (DFS) will be the primary end-point of efficacy in this Phase III trial. It will be measured from the date of randomization to the date of progression or death, whatever the cause.
  Overall Survival will be also evaluated and it is defined as the time from the date of randomization to the date of death from any cause or to the date of last follow-up.

SECONDARY OUTCOMES:
Evaluation of Vitamin D receptors and 25(OH)D by Breslow thickness. | baseline and after 1 year of treatment
  Evaluation at baseline of Vitamin D receptors and 25(OH)D by Breslow thickness. Change in time of 25(OH)D serum level by VDR and other genes involved in vitamin D metabolisms.
  Percentages of patients at desired levels of 25(OH)D (30 ng/ml) during 1 year. Toxicity.
  Compliance. OS.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Testori, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy